CLINICAL TRIAL: NCT00212277
Title: Phase3,Open-label,Long-term,NSAID-Add-on,Clinical Trial of Mono-phase Low-dose Oral Contraceptive Pill for Treatment of Dysmenorrhea Associated With Endometriosis.
Brief Title: Efficacy and Safety,Long-term Study of Low-dose Oral Contraceptive Pill to Treat Dysmenorrhea.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nobelpharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IKH-01-5
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2010-09-10 (Estimated); Status verified 2010-09

CONDITIONS: Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea | interventions — ovcon 35

INTERVENTIONS:
Drug: Norethindrone,Ethinyl Estradiol

SUMMARY:
The purpose of this long-term study is to determine whether combination oral contraceptive pill of Norethindrone & Ethinyl estradiol is effective in the treatmentof dysmenorrhea associated with endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* dysmenorrhea associated with endometriosis

Exclusion Criteria:

* severe hepatopathy
* pregnant woman

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-02; Primary Completion 2006-09 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naoki Terakawa, M.D.,Ph.D., Study Director — Tottori University,Tottori,Japan